CLINICAL TRIAL: NCT03654950
Title: PEPP - Patient Empowerment With the Patient Perspective
Brief Title: Patient Empowerment With the Patient Perspective
Acronym: PEPP
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Högskolan Väst (Unknown)
Responsible Party: Principal Investigator, Eva Angenete, Associate professor, consultant surgeon, Sahlgrenska University Hospital
Other Study IDs: PEPP
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Interviews and questionnaires

SUMMARY:
The overall aim with this study is to gain a deeper understanding of patient perceptions regarding empowerment in relation to a health platform.

DETAILED DESCRIPTION:
This is a two-stage study design. The first stage consists of focus groups interviews. Three focus groups with 6-8 patients (colorectal cancer patients diagnosed at least one year ago) in each group, will be invited. The focus group interviews will be moderated by one researcher, but accompanied with a second observing researcher. The participants will be identified using the regional Swedish ColoRectal Cancer Registry in Västra Götaland. The participants will be contacted by a short letter (appendix) indicating that we will call them with more information. The participants will by phone be asked to participate in the study and then invited to the focus groups.

The second phase of the project includes a questionnaire, which will be sent to 200 patients from the same population. The questionnaires will be delivered by using the Sunet Survey system, which is a system approved by University of Gothenburg. If the participants prefers a paper copy, or lack the possibility to reply online, a paper copy will be send via mail instead.

At this moment the investigators have developed a questionnaire, which may be refined due to the understating achieved from the focus group interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patient with colorectal cancer

Exclusion Criteria:

* Inability to give informed consent or speaking and reading the Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Patient reported experiences in themes | 1 day
  interview

SECONDARY OUTCOMES:
Patient reported experiences divided into themes | 12 months
  Interview

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, Principal Investigator — Sahlgrenska University Hospital and University of Gothenburg
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided